

Document Date: 8/29/2024

# **Human Subjects Informed Consent Form**

Idaho State University Department of Dental Hygiene

The Impact of Barre Stretching on Self-Reported Stress and Pain Levels Among Entry-Level
Dental Hygiene Students

Vanessa Whiley, RDH, BS, MS(c)

### What is the Research?

You have been asked to participate in a 6-week study that researches whether a relationship exists between a Barre stretching and breathing intervention and the self-reported stress and pain levels among entry-level dental hygiene students. The Human Subjects Committee at Idaho State University has evaluated this research project, IRB Number: IRB-FY2024-106.

#### **Procedures**

If you agree to participate in this study, you agree to the following procedures:

- Upon agreeing to participate, an informed consent document will be signed and returned to the investigator, and you will receive a copy.
- After the researcher has qualified you to participate, you will be randomly selected to an experimental group to receive the intervention being tested or selected to a control group.
- Record your stress level on the Perceived Stress Scale (PSS-10) pre-intervention.
- Record your pain level on the Numerical Pain Rating Scale/Visual Analog Scale (NPRS/VAS-11) scale pre-intervention.
- Experimental Group: Complete two (2) 15-minute Barre stretching video exercises weekly (Monday and Thursday).
- Record your stress level on the Perceived Stress Scale (PSS-10) post-intervention.
- Record your pain level on the Numerical Pain Rating Scale/Visual Analog Scale (NPRS/VAS-11) scale post-intervention.
- A copy of the results of the study will be sent to participants upon request. Data will be reported in group format with no personal identifiers.

## **Voluntary Participation**

This study is voluntary—you do not have to take part if you do not want to. You may leave the study at any time and for any reason. Participation in this study will not affect any dental hygiene treatment provided at the clinic.

#### **Risks and Benefits**

Despite all attempts to preserve privacy and anonymity, there may be a slight risk of your identity being recognized, however, all data on the pre-test and post-test will be de-identified. Participants will be asked to enter the last four digits of their phone number to link the pre-test to the post-test. Once data has been collected and entered on a spreadsheet, the last four digits of the phone number will be removed.

There are no personal benefits for taking part in this research. However, the information gained from this study may help researchers learn more about a treatment modality that may reduce selfreported stress and pain levels among entry-level dental hygiene students, and lower MSD risk.

# **Privacy and Confidentiality**

To protect your confidentiality, all personal identifiers will be destroyed once data is collected from the daily journal. Data collected from this study will be uploaded into Box which is a HIPPA certified electronic storage tool at Idaho State University. Box is password protected and has firewall protection. Only the principal investigator and co investigators will have access to the data collected from the study. The data will be stored and secured in Box for seven years, at that point all material of the study will be destroyed by Idaho State University following university protocol.

## Questions

If you have any additional questions about the study, you may contact the primary investigator.

## **Primary Investigator**

Vanessa Whiley, RDH, BSDH, MSDH (c) vanessawhiley@isu.edu

### **Faculty Thesis Co-Chairpersons**

Leciel Bono, RDH-ER, MS Graduate Program Director Idaho State University Mail Stop 8048 Pocatello, ID 83209

Email: bonoleci@isu.edu

Phone: (208) 242-8158

Crystal Kanderis Lane, RDH, MS **Assistant Professor** Idaho State University Mail Stop 8048 Pocatello, ID 83209

Email: crystalkanderislane@isu.edu

Phone: (208)-240-4209

I have read the information in the consent form. I have been given an opportunity to ask questions, and any questions I had have been answered to my satisfaction. I have been given a copy of the informed consent.

I give my consent for the results of the pilot study to be published or discussed using my photos and journal. No information will be included that will reveal my identity.

I HAVE REVIEWED THIS CONSENT FORM AND UNDERSTAND AND AGREE TO ITS CONTENTS.

| Printed Name | Signature | Date |
|--------------|-----------|------|